CLINICAL TRIAL: NCT05478993
Title: A Phase 2 Study of Selinexor, Pomalidomide, and Dexamethasone For Multiple Myeloma With Central Nervous System Involvement
Brief Title: Selinexor, Pomalidomide, and Dexamethasone For Multiple Myeloma With CNS Involvement
Acronym: SPODUMENE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Qingdao Municipal Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, MD, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01/20/2022
Record Dates: First submitted 2022-07-24; First posted 2022-07-28 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Multiple Myeloma
Keywords: Central Nervous System
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with multiple myeloma with CNS involvement to receive Selinexor (60 mg QW), pomalidomide (4 mg/day, on Days 1-21), and dexamethasone (40 mg/day, on Days 1, 8, 15, 22), with all agents dosed 28 days per cycle.
  If patients reach maximum efficacy and have received SPD treatment for 8-12 cycles, maintenance treatment of Selinexor (20-60mg QW, optimal dose determined by the investigator) will be started and continued until disease progression or intolerable adverse events.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Selinexor, pomalidomide and dexamethasone (Experimental): Patients diagnosed with multiple myeloma with CNS involvement to receive SPD treatment.
  Interventions: Drug: SPD：Selinexor Oral Tablet, Pomalidomide, Dexamethasone

INTERVENTIONS:
Drug: SPD：Selinexor Oral Tablet, Pomalidomide, Dexamethasone — Patients diagnosed with multiple myeloma with CNS involvement to receive Selinexor (60 mg QW), pomalidomide (4 mg/day, on Days 1-21), and dexamethasone (40 mg/day, on Days 1, 8, 15, 22), with all agents dosed 28 days per cycle.
  If patients reach maximum efficacy and have received SPD treatment for 8-12 cycles, maintenance treatment of Selinexor (20-60mg QW, optimal dose determined by the investigator) will be started and continued until disease progression or intolerable adverse events.

SUMMARY:
This is a single-arm, open-label, multicenter, exploratory study initiated by investigator to evaluate the efficacy and safety of Selinexor (S) combined with pomalidomide (P) and dexamethasone (D) in the treatment of multiple myeloma with CNS involvement.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter, exploratory study. The study plans to enroll patients diagnosed with multiple myeloma with CNS involvement to receive Selinexor (60 mg QW), pomalidomide (4 mg/day, on Days 1-21), and dexamethasone (40 mg/day, on Days 1, 8, 15, 22), with all agents dosed 28 days per cycle.

If patients reach maximum efficacy and have received SPD treatment for 8-12 cycles, maintenance treatment of Selinexor (20-60mg QW, optimal dose determined by the investigator) will be started and continued until disease progression or intolerable adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients with multiple myeloma with measurable lesions as assessed using the updated International Myeloma Working Group Response Criteria.
3. Multiple myeloma patients with central nervous system involvement (CNS-MM): the presence of plasma cells in the cerebrospinal fluid (CSF), and/or leptomeningeal, dural, or intraparenchymal involvement as assessed using imaging modalities (MRI, CT or PET-CT), and/or tissue biopsy; or eye involvement confirmed by ophthalmologists, with or without neurological symptoms.
4. ECOG ≤ 2, with expected survival of more than 3 months.
5. No active infectious diseases.
6. Major organs without serious organic diseases (except renal insufficiency caused by multiple myeloma).
7. Female patients are not during pregnancy or breastfeeding; fertile men or women agree to use appropriate methods of contraception 4 weeks before study treatment, during treatment and drug suspension, and within 4 weeks after the end of study treatment.
8. Be able to cooperate with study follow-up. Patients understand the disease characteristics and voluntarily join this study to receive treatments and study follow-ups.
9. Have signed informed consent. Informed consent was signed by the patient or by an immediate family member. Considering the patient 's condition, if the patient' s signature is unfavorable for disease treatment, the informed consent form should be signed by the legal guardian or the patient 's immediate family member.

Exclusion Criteria:

1. Patients with active hepatitis B (HBV), hepatitis C (HCV), and other acquired, congenital immunodeficiency diseases;
2. According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) 5.0, baseline with grade 2 or higher peripheral neuropathy or neuralgia;
3. Severe thrombotic events before treatment;
4. Patients with uncontrolled or severe cardiovascular disease, including myocardial infarction within 6 months before enrollment, New York Heart Association (NYHA) defined grade III-IV heart failure, uncontrolled angina pectoris, clinically significant pericardial disease or cardiac amyloidosis;
5. Major surgery within 30 days before enrollment;
6. Epilepsy and dementia which requires drug treatment, and other mental disorders which cannot understand or follow the study protocol;
7. According to the protocol or the investigator 's judgment, any severe physical illness or mental illness may interfere with participation in this clinical study;
8. Drug abuse, medical, psychological or social conditions that may interfere with the participation of subjects in the study or evaluation of study results;
9. Patients who are receiving other experimental treatment;
10. Pregnant or lactating women;
11. Not suitable for enrollment per investigators' judgements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Assessed using the updated International Myeloma Working Group Response Criteria

SECONDARY OUTCOMES:
Overall survival | From date of enrollment until date of death from any cause, assessed up to 24 months.
  Assessed using the updated International Myeloma Working Group Response Criteria
Overall response rate | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Assessed using the updated International Myeloma Working Group Response Criteria
Adverse Events | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Assessed using the CTCAE criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, M.D., Principal Investigator — Peking University People's Hospital
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Qingdao Municipal Hospital, Qingdao, Shandong

IPD SHARING:
Plan to Share IPD: No